CLINICAL TRIAL: NCT03432793
Title: A Phase 1, Fixed-Sequence, Open-Label Drug-Drug Interaction Study to Assess the Effect of Fluvoxamine (CYP1A2 Inhibitor), Cigarette Smoking (CYP1A2 Inducer) and Itraconazole (CYP3A4 Inhibitor) on the Pharmacokinetics of TD-9855 in Healthy Subjects
Brief Title: Drug-Drug Interaction (DDI) Study for TD-9855
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0172
Record Dates: First submitted 2018-02-02; First posted 2018-02-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Drug Drug Interaction (DDI)
Keywords: DDI; Itraconazole; Fluvoxamine; TD-9855; Smoking; Caffeine; CYP1A2; CYP3A4
MeSH Terms: conditions — Smoking | interventions — ampreloxetine; Fluvoxamine; Itraconazole; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TD-9855 + Fluvoxamine + Caffeine (Experimental): Male smokers will receive TD-9855, fluvoxamine, and caffeine
  Interventions: Drug: TD-9855; Drug: Fluvoxamine; Drug: Caffeine
- TD-9855 + Itraconazole + Caffeine (Experimental): Male non-smokers will receive TD-9855, itraconazole, and caffeine
  Interventions: Drug: TD-9855; Drug: Itraconazole; Drug: Caffeine

INTERVENTIONS:
Drug: TD-9855 — oral tablet, QD
Drug: Fluvoxamine — oral tablet, QD
  Arms: TD-9855 + Fluvoxamine + Caffeine
Drug: Itraconazole — oral tablet solution, QD
  Arms: TD-9855 + Itraconazole + Caffeine
Drug: Caffeine — oral solution, single dose

SUMMARY:
This study is designed to assess the effect of fluvoxamine, itraconazole and smoking on the PK disposition of multiple doses TD-9855 in healthy male subjects. The study will also assess the relationship between caffeine PK and TD-9855 PK disposition in healthy male smokers and non-smokers.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written, signed informed consent
* Male subjects 19 to 55 years of age (inclusive)
* Body mass index 19 to 32 kg/m2 (inclusive), and weigh at least 55 kg
* No clinically important abnormal physical findings as determined by the Principal Investigator (PI) at the screening and Day -1 examinations
* Negative for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV) antibody at screening.
* No clinically important laboratory abnormalities as determined by the PI
* Ability to communicate effectively with the Investigator and to comply with all study requirements, restrictions, and direction of the clinic staff
* Male subjects must abstain from sexual intercourse or use a highly effective method of birth control
* Male smokers: Subjects who self-report to have smoked > 9 cigarettes per day for at least 6 month prior to screening as confirmed by urine cotinine test at screening and Day -1.
* Male smokers: Subjects must be willing to continue consistent use of their tobacco products throughout the study.
* Additional inclusion criteria apply

Exclusion Criteria:

* Positive for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV) antibody at screening.
* History or presence of clinically significant respiratory, gastrointestinal, renal, hepatic, hematologic, neurologic (including history of seizure and insomnia), cardiovascular (including postural orthostatic hypotension or tachycardia), psychiatric (including depression and known addictive disorders), musculoskeletal, genitourinary (including urinary retention), immunologic, or dermatologic disorder.
* Any other condition that, in the opinion of the PI, would confound or interfere with study participation; evaluation of safety, tolerability, or PK of the investigational drug; or prevent compliance with the study protocol
* Any history of suicide attempts/ideation or current suicidal ideation.
* Have participated in another clinical trial of an investigational drug (or medical device) within 30 days (or 5 half-lives of the investigational drug if longer than 30 days) prior to Screening, or are currently participating in another trial of an investigational drug (or medical device), or intending to participate in another trial of an investigational drug (or medical device) before completion of all scheduled safety evaluations in this trial
* Additional inclusion criteria apply

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-04-21 (Actual); Study Completion 2018-04-21 (Actual)

PRIMARY OUTCOMES:
Change in TD-9855 plasma exposure when administered with itraconazole or fluvoxamine | Day 9 and Day 24

SECONDARY OUTCOMES:
Correlation between caffeine PK disposition and TD-9855 plasma exposure | Day 9 and Day 24
  Correlation co-efficient will be calculated between caffeine/paraxanthine ratio at 4hr after caffeine dose and TD-9855 plasma AUC on Day 9 and Day 24.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.